CLINICAL TRIAL: NCT07400393
Title: Healey ALS MyMatch Common Screening Protocol (MCSP) for Determining Preliminary Eligibility for ALS MyMatch Early Phase Clinical Trials
Brief Title: Healey ALS MyMatch Common Screening Protocol
Acronym: MCSP
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Suma Babu, Associate Professor of Neurology at Harvard Medical School and Co-Director of the Neurological Clinical Research Institute (NCRI), Massachusetts General Hospital
Other Study IDs: 2025P002080
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: ALS; ALS (Amyotrophic Lateral Sclerosis); ALS - Amyotrophic Lateral Sclerosis
Keywords: ALS; Amyotrophic Lateral Sclerosis; MyMatch; ALS MyMatch; MyMatch Program; MCSP; MyMatch Common Screening Protocol; Early Phase; Biomarker; Phase I; Phase II; Healey; NCRI; ALS Trials; MGB
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 45 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of the Healey ALS MyMatch Common Screening Protocol (MCSP), an observational study, is to identify individuals with ALS who may be eligible to be matched to a currently enrolling ALS MyMatch trial. Participants will complete a MCSP Screening Visit and undergo clinical assessments, laboratory testing, and biomarker analyses to determine preliminary trial eligibility. The study also characterizes clinical, genetic, and biofluid biomarker profiles, assesses the prevalence of ALS-associated gene variants, and banks blood samples for future ALS and biomarker research. MCSP enables simultaneous screening for multiple trial-specific biomarkers and uses a targeted medical history form to optimize matching of participants to appropriate MyMatch trials.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Adults > 18 years of age.
3. Diagnosis of symptomatic ALS that meets either the revised El Escorial Criteria.(clinically possible, probable, probable lab-supported, or definite) or the Gold Coast Criteria.
4. Available or pending clinically obtained CLIA ALS genetic panel report.
5. Time since onset of weakness due to ALS ≤ 24 months at the time of MCSP screening.
6. Slow VC ≥ 65% of predicted capacity value for gender, height and age at screening.
7. Clinically unremarkable Complete Blood Counts as per SI's discretion, including but not limited to Hemoglobin ≥ 9 g/dL.
8. Ability and willingness to complete all study procedures per SI's assessment.
9. Negative pregnancy test at screening for women of child-bearing potential (WOCB), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months).

Exclusion Criteria:

1. Clinically significant unstable medical or surgical condition that would pose a risk to the participant's trial procedural participation or interfere with data collection, per SI's assessment.
2. Presence of cognitive or mental health disorders impairing ability to provide informed consent for the study per SI assessment.
3. Active cancer or history of cancer, unless it was successfully treated for durable remission or cure more than 3 years ago. (Note that basal cell carcinoma, squamous cell carcinoma in situ, cervical carcinoma in situ, prostatic carcinoma in situ, or other malignancies that have been curatively excised at any time previously and with no evidence of disease recurrence for at least 3 years are not exclusionary.)
4. Prior solid organ transplantation.
5. Use of investigational treatments for ALS (off-label use or active participation in a clinical trial) within 5 half-lives (if known) or 30 days (whichever is longer) prior to the MCSP Screening Visit. (Please refer to the Manual of Procedures (MOP) for current list of experimental therapies)
6. Screening 12-lead ECG showing QT interval corrected for rate (QTcF) > 470 msec for women and > 450 msec for men, absence of second degree or higher AV block or other clinically significant cardiac arrythmias.
7. Clinically significant abnormalities in the Comprehensive Metabolic Panel per SI's assessment, including but not limited to:

   1. Serum alanine aminotransferase or aspartate aminotransferase > 3 times the upper limit of normal, or serum bilirubin > 1.5 × upper limit of normal
   2. Estimated GFR (eGFR) of < 30 mL/min/1.73m2
8. Other clinically significant electrolyte and metabolic abnormalities
9. If female, breastfeeding, pregnant, or of child-bearing potential and unwilling to use effective contraception for duration of the trial and after discontinuing treatment as outlined in the ALS MyMatch trial protocol.
10. Clinically significant unstable medical conditions (other than ALS) that would pose a risk to the participant, per SI's assessment (e.g., cardiovascular instability, systemic infection,), or clinically significant laboratory abnormality or ECG changes.
11. Exposure at any time to any gene therapies under investigation for the treatment of ALS (off-label use or investigational).
12. Participants who require Permanent assisted ventilation (PAV). PAV defined as more than 22 hours per day of noninvasive or invasive mechanical ventilation for more than seven consecutive days. The date of onset of PAV is the first day of the seven days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target populations for MCSP and ALS MyMatch trials will initially focus on subgroups of individuals with ALS, including those with early-stage disease. Some ALS MyMatch trials will further target those with specific biomarkers or genetic markers for inclusion in a specific trial.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-03-16 (Estimated); Primary Completion 2029-03-16 (Estimated); Study Completion 2029-03-16 (Estimated)

PRIMARY OUTCOMES:
Preliminary eligibility to be matched to a MyMatch Trial | From enrollment to the end of the 45-day MCSP screening period or at the end of completing a baseline visit for a MyMatch trial.
  To determine preliminary eligibility of early ALS (< 24 months from weakness onset) participants for actively enrolling ALS MyMatch trial(s)

SECONDARY OUTCOMES:
Repository for future research | From enrollment to the end of the 45-day MCSP screening period or at the end of completing a baseline visit for a MyMatch trial. Samples will be banked indefinitely for future research on ALS and related diseases.
  To build an ALS biofluid, genetic and data repository for future clinical and translational research.
Prevalence of gene mutations | From enrollment to the end of the 45-day MCSP screening period or at the end of completing a baseline visit for a MyMatch trial. Samples will be banked indefinitely for future research on ALS and related diseases.
  To characterize the prevalence of participants with causative or risk modifier gene mutations in the MCSP
Collect and bank samples | From enrollment to the end of the 45-day MCSP screening period or at the end of completing a baseline visit for a MyMatch trial. Samples will be banked indefinitely for future research on ALS and related diseases.
  To collect and bank blood samples for future biofluid biomarker analyses